CLINICAL TRIAL: NCT06787963
Title: Quantitative Proteomic Analysis of Minor Whey Proteins and Peptides of Human Milk Across Five Neonatal Groups Classified by Birth Weight During the Three Stages of Lactation
Brief Title: Exploring Minor Proteins and Peptides in Human Milk: a Proteomic Analysis Across Lactation Stages
Acronym: PROTEOM-MILK
Status: Recruiting | Type: Observational
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Hospital Universitario Reina Sofia de Cordoba (Other Government); Universidad de Granada (Other); Universidad de Córdoba (Other)
Responsible Party: Sponsor
Other Study IDs: PROTEOM-MILK
Record Dates: First submitted 2025-01-08; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Low Birthweight Infant; Preterm; Very Low Birth Weight Preterms
Keywords: low birth weight; prematurity; gestational age; human milk; bioactive peptides; proteomics; lactation; whey protein
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human milk samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- 30 extremely low birth weight: extremely low birth weight (< 1000 g)
- 30 very low birth weight: very low birth weight (1000-1499g)
- 30 low birth weight: low birth weight (1500-2499g)
- 30 adequate birth weight: adequate birth weight (2500-3999g)
- 30 high birth weight: high birth weight (4000g or >)

SUMMARY:
Human milk (HM) is the optimal food source for the nutrition, growth, and development of newborns. The protein fraction of HM plays a crucial role in the healthy development of infants. HM contains a wide variety of minor whey proteins and peptides with important bioactive functions, many of which are still unknown. Proteomics allows for the study of biological samples with inherently complex protein mixtures. Proteins are essential for the development of living organisms, both in quantitative and qualitative terms. The combination of proteomic techniques currently enables the study of protein variability and minor peptides in HM across different lactation stages and allows for differential quantification according to gestational age and birth weight. However, studies on the human milk serum proteome during these stages are limited. The aim is to explore the minor whey proteins and peptides in human milk through a longitudinal analysis of five groups of breastfeeding mothers (with 30 extremely low birth weight newborns, 30 very low birth weight newborns, 30 low birth weight newborns, 30 adequate birth weight newborns, and 30 high birth weight newborns). Gestational age will also be considered to ensure homogeneous group distribution according to this condition. HM samples will be collected from each mother during three lactation periods after birth: within the first 48 hours (colostrum), at 5-14 days (transitional milk), and at 100-120 days (mature milk) for the five birth weight groups. In these neonatal/infant groups, minor proteins from whey fraction and peptides will be separated, quantified, and identified using label-free proteomic techniques. This study aims to expand our understanding of the minor proteins and peptides in human milk and their bioactive roles in neonatal health. By examining these components across different birth weight groups and lactation stages, the research will offer insights into how protein and peptide profiles vary by gestational age and birth weight, potentially influencing neonatal development. The findings from this proteomic analysis could not only demonstrate the complexity of human milk composition but also contribute to targeted nutritional support for preterm or low-birth-weight infants, customizing protein supplementation in HM banks and therefore enhancing their growth and developmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy mothers
* With monitored pregnancies within the care area of the Reina Sofía University Hospital in Córdoba
* With newborns expected to be exclusively breastfed until 4 months

Exclusion Criteria:

* Mothers whose newborns have any of the following conditions: congenital malformation, chromosomal abnormality, hypoxia-ischemia, gastroschisis, polycythemia, hypoglycemia, sepsis, blood incompatibility
* Pathological pregnancy, pregnancy by in vitro fertilization, or multiple pregnancies
* With no plan to exclusively breastfeed until 4 months
* Under medical treatment
* Have a drug addiction
* Refuse informed consent
* Have had previous breast surgery
* Live outside the metropolitan area

Ages: 0 Days to 120 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Five groups of breastfeeding mothers: Group 1 (n=30) - with neonates of extremely low birth weight; Group 2 (n=30) - with neonates of very low birth weight; Group 3 (n=30) - with neonates of low birth weight; Group 4 (n=30) - with neonates of adequate birth weight; Group 5 (n=30) - with neonates of high birth weight. Additionally, gestational age will be considered to achieve a homogeneous distribution of the groups according to this condition.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Minor whey proteins: Lysozyme | Human Milk collection after birth - Time 1: at 48 hours (colostrum),Time 2: at 5-14 days (transitional milk), Time 3: at 100-120 days (mature milk)
  Concentration of lysozyme in ng/ml will be measured using immunoassays (Enzyme-Linked ImmunoSorbent Assay).
Minor whey proteins: Lactoferrin | Human Milk collection after birth - Time 1: at 48 hours (colostrum),Time 2: at 5-14 days (transitional milk), Time 3: at 100-120 days (mature milk)
  Concentration of lactoferrin in mg/ml will be measured using immunoassays (Enzyme-Linked ImmunoSorbent Assay).
Minor whey proteins: Bile salt-dependent lipase (BSDL) | Human Milk collection after birth - Time 1: at 48 hours (colostrum),Time 2: at 5-14 days (transitional milk), Time 3: at 100-120 days (mature milk)
  Concentration of bile salt-dependent lipase (BSDL) in µg/ml will be measured using immunoassays (Enzyme-Linked ImmunoSorbent Assay).
Minor whey proteins: Lactoperoxidase | Human Milk collection after birth - Time 1: at 48 hours (colostrum),Time 2: at 5-14 days (transitional milk), Time 3: at 100-120 days (mature milk)
  Concentration of lactoperoxidase in ng/ml will be measured using immunoassays (Enzyme-Linked ImmunoSorbent Assay).
Minor whey proteins: Alpha-1-antitrypsin | Human Milk collection after birth - Time 1: at 48 hours (colostrum),Time 2: at 5-14 days (transitional milk), Time 3: at 100-120 days (mature milk)
  Concentration of alpha-1-antitrypsin in ng/ml will be measured using immunoassays (Enzyme-Linked ImmunoSorbent Assay).
Proteome | Human Milk collection after birth - Time 1: at 48 hours (colostrum),Time 2: at 5-14 days (transitional milk), Time 3: at 100-120 days (mature milk)
  Protein signatures will be assessed through a proteomic analysis using nano-liquid chromatography (nESI-MS/MS). The analysis will be followed by bioinformatic analysis with dedicated software to analyze and achieve the relative quantification of differential proteins. A specific database representing the human proteome, updated in the UNIPROT repository, will be used. The results will be compared against the protein databases available in international platforms such as SWISS-Prot, NCBI, EBI, and TrEMBL. The results are typically expressed in units or formats that reflect the relative abundance or quantitative values of proteins or peptides, such as spectral counts, percentage and µg/ml.
Free peptides, primarily derived from β-casein | Human Milk collection after birth - Time 1: at 48 hours (colostrum),Time 2: at 5-14 days (transitional milk), Time 3: at 100-120 days (mature milk)
  Free peptides will be expressed in counts per peptide. Human milk samples will undergo trypsin digestion prior to analysis by liquid chromatography-mass spectrometry (LC-MS).

SECONDARY OUTCOMES:
Muscular ecography | After birth - Time 1: at 48 hours,Time 2: at 5-14 days, Time 3: at 100-120 days
  Muscle thickness will be measured using a Phillips HD ultrasound equipment, with a high-frequency linear probe (7.5 MHz - 15 MHz), in B-mode. The thickness (expressed in mm) of the right quadriceps muscle and subcutaneous tissue will be measured, taken at the midpoint between the greater trochanter and tibial plateau: one anteroposterior in longitudinal section, another anteroposterior in transverse plane, and another perpendicular to the latter in the same plane.
Transfontanellar ecography | After birth - Time 1: at 48 hours,Time 2: at 5-14 days, Time 3: at 100-120 days
  Brain structure and anatomy will be measured using a convex probe with a frequency range of (3.5 - 7 MHz) in B-mode. Longitudinal and transverse sections will be measured, and the thickness of the frontal cortex and the maximum thickness of the corpus callosum will be measured in millimeters (mm).

OTHER OUTCOMES:
General information - Mothers | After birth - Time 1: at 48 hours,Time 2: at 5-14 days, Time 3: at 100-120 days (mothers will be asked if any changes have occurred)
  Mothers will complete a general questionnaire to gather information on sociodemographic factors, pregnancy, breastfeeding, medical conditions or complications, medications, and lifestyle habits
General information - Newborns | After birth - Time 1: at 48 hours,Time 2: at 5-14 days, Time 3: at 100-120 days (mothers will be asked if any changes have occurred)
  A general questionnaire will be completed regarding newborn characteristics, including gestational age, birth weight and length, sex, feeding type, and any pre- and/or postnatal complications or infections.
Dietary intake and eating habits | After birth - Time 1: at 48 hours,Time 2: at 5-14 days, Time 3: at 100-120 days
  Food Consumption Frequency Questionnaire (CFCA) at the beginning of the study will be conducted, along with a 3-day food diary during the three stages of breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Gómez-Chaparro Moreno, MD, Ph.D, Principal Investigator — Maimonides Biomedical Research Institute of Cordoba (IMIBIC)
Locations (2):
- Spain (2):
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Maimonides Biomedical Research Institute of Cordoba (IMIBIC), Córdoba, Córdoba

IPD SHARING:
Plan to Share IPD: No
The datasets generated and analyzed in this study are not publicly available due to data regulations and ethical considerations. Participants consented to the use of their data exclusively by the original team of investigators, ensuring their privacy and adherence to consent agreements.